CLINICAL TRIAL: NCT00314184
Title: Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled Phase 3 Study of the Efficacy and Safety of Quetiapine Fumarate and Lithium as Monotherapy for up to 104 Weeks Maintenance Treatment of Bipolar I Disorder in Adult Patients
Brief Title: Quetiapine Fumarate Bipolar Maintenance Monotherapy
Acronym: SPaRCLe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1447C00144; EUDRACT 2004-000915-25
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2008-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I disorder.
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: quetiapine fumarate
  Other Names: Seroquel

SUMMARY:
This is a multicenter, randomized, parallel-group, double-blind, placebo-controlled study to evaluate the efficacy and safety of quetiapine and lithium (comparator in the study) for up to 104 weeks of maintenance treatment in adult patients with Bipolar I Disorder.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 18 years or older
* A diagnosis of Bipolar I Disorder
* Have a current manic, depressed or mixed episode
* Have had a manic, depressed or mixed episode during the last 26 weeks that was treated with quetiapine
* Female patients of childbearing potential must be using a reliable method of contraception

Exclusion Criteria:

* Pregnancy
* Substance or alcohol dependence at enrollment
* Unstable thyroid function
* Unstable Diabetes
* Unstable or inadequately treated medical illness e.g., angina pectoris and hypertension
* Use of an experimental drug within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1255 (Actual)
Dates: Start 2005-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Time from randomization to recurrence of a mood event

SECONDARY OUTCOMES:
Time from randomization to recurrence of a manic event
Time from randomization to recurrence of a depressed event

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca CNS Medical Science Director, MD, Study Director — AstraZeneca
Locations (95):
- United States (30):
  - Research Site, Cerritos, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, North Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Terre Haute, Indiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Flowood, Mississippi
  - Research Site, Saint Charles, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Clementon, New Jersey
  - Research Site, Rochester, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Portland, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Lake Jackson, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Seattle, Washington
- Argentina (6):
  - Research Site, Capital Federal
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Lanús
  - Research Site, Mendoza
  - Research Site, Rosario
- Bulgaria (3):
  - Research Site, Burgas
  - Research Site, Plovdiv
  - Research Site, Sofia
- Colombia (4):
  - Research Site, Antioquia
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Pereira
- India (10):
  - Research Site, Ahmedabad
  - Research Site, Chennai
  - Research Site, Jaipur
  - Research Site, Kanpur
  - Research Site, Lucknow
  - Research Site, Mangalore
  - Research Site, Manipal
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Visakhapatnam
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Sarawak
- Mexico (3):
  - Research Site, León
  - Research Site, México
  - Research Site, San Luis Potosí City
- Research Site, Lima, Peru
- Philippines (5):
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Mandaluyong
  - Research Site, Manila
  - Research Site, Quezon City
- Romania (12):
  - Research Site, Arad
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Com Jebel
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Piteşti
  - Research Site, Sibiu
  - Research Site, Târgovişte
  - Research Site, Târgu Mureş
- Russia (3):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Taiwan (4):
  - Research Site, Kaohsiung Hsien
  - Research Site, Taipei
  - Research Site, Taoyuan
  - Research Site, Taoyuan Hsien
- Research Site, Bangkok, Thailand
- Ukraine (8):
  - Research Site, Dnipro
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Simferopol
  - Research Site, Vinnitsa

REFERENCES:
- [Derived] Weisler RH, Nolen WA, Neijber A, Hellqvist A, Paulsson B; Trial 144 Study Investigators. Continuation of quetiapine versus switching to placebo or lithium for maintenance treatment of bipolar I disorder (Trial 144: a randomized controlled study). J Clin Psychiatry. 2011 Nov;72(11):1452-64. doi: 10.4088/JCP.11m06878. PMID 22054050